CLINICAL TRIAL: NCT01623726
Title: Transcranial Direct Current Stimulation (tDCS) as Therapeutical Strategy for Negative Symptoms in Schizophrenia: a Double-blind Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) as Therapeutical Strategy for Negative Symptoms in Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: To be submitted for grant application
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Brunoni, Prof. Dr., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAISM-001
Record Dates: First submitted 2012-06-08; First posted 2012-06-20 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Transcranial Direct Current Stimulation; Schizophrenia
Keywords: Transcranial Direct Current Stimulation; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS active (Experimental): Active tDCS as foreseen in research protocol: daily sessions for 10 days with 2mA intensity stimulation during 20 minutes.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- tDCS sham (Placebo Comparator): Sham tDCS : as foreseen in research protocol: sham stimulation with initial stimulation followed by turning off the device during the same time of intervention as to guarantee blinding
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation. Daily sessions with a total of 10 days intervention. Each intervention will take place with a 2mA intensity during 20 minutes. The current will be delivered by "Chattanooga Iontophoresis Dual Channel Delivery Device", that stands for a 2-channels tDCS device in which previous dosage can be set as default to maintain frequently used treatment parameters. Main features include (a) Beeping alerts if electrode fault for open current or high impedance, low battery, treatment completion or power left on; (b)automatic 30 second current ramp up and down during power on/off keeps patient comfortable; (c) Current can be set in 0.1 mA increments between 0.5 mA and 4 mA.

SUMMARY:
The current research is aimed at using Transcranial Direct Current Stimulation (tDCS) as complementary therapeutic tool in the treatment of schizophrenia. Patients will be randomized into two groups (tDCS-active x tDCS-sham) accordingly to detailed protocol. Main outcome will be measured by specific clinical rating scales based on the assessment of negative symptoms. A total of 40 patients ought to be enrolled as specified in methodology. Secondary outcomes shall include collateral effects evaluation, anxiety and depressive scales as well as clinical monitoring.

DETAILED DESCRIPTION:
Overview

The present study is a double-blind randomized clinical trial in which patients should be allocated from a General Psychiatry Service into two groups (tDCS-active x tDCS-sham). Subjects who fulfilled eligibility criteria will undergo ten days of consecutive stimulation (active or sham) and will return after two to four weeks for final clinical assessment. Patients who shown no response in rating scales and that were allocated to sham intervention group will be able to choose whether or not they want to undergo the active intervention at follow up (partial cross-over)

ELIGIBILITY:
Inclusion Criteria:

* patients with age between 18-59 years
* diagnostic of Schizophrenia or Schizoaffective Disorder as stated by DSM-IV and confirmed by SCID (Structured Clinical Interview for DSMIV), to be tested by a psychiatrist
* baseline score higher than 20 for negative symptoms at PAAN
* patients able to read and understand Portuguese.

Exclusion Criteria:

* other psychiatric diagnosis
* criteria for bipolar disorder; dementia; other psychotic disturbs; substance related disorders
* presence of other severe neurological or clinical diseases
* presence of suicidal behavior (planning or attempt in the previous 4 weeks)
* pregnancy
* incapacity of coping with the informed consent
* specific tDCS limitations (such as anatomic problems)

Regarding medication: all patients should have stable dosology of medications for at least 6 weeks

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Negative Symptoms Rates as assessed by the PAANS | Assessment at 0(baseline), 2 weeks and 4 weeks (final outcome) - Positive and Negative Syndrome Scale (PAANS)
  Comparison between follow u and baseline PAANS scores with emphasis in negative symptoms scores

SECONDARY OUTCOMES:
Mental Mini Exam | Assessment at 0(baseline), 2 weeks and 4 weeks (final outcome) - Cognitive Screening assessment as performed by the Mental Mini Exam
  cognitive evaluation as assessed by the Mental Mini Exam
Moca rating Scale | Assessment at 0(baseline), 2 weeks and 4 weeks (final outcome) - Cognitive assessment by MoCa Test
  comparison between follow up and baseline scores in Cognitive evaluation as assessed by MoCa Test
Stroop Victoria | Assessment at 0(baseline), 2 weeks and 4 weeks (final outcome) - Cognitive assessment by Stroop - Victoria version
  comparison between follow up and baseline scores in atention and inhibitory control as assessed by Stroop Victoria
Neuropsychological Assessment | Assessment at 0(baseline), 2 weeks and 4 weeks (final outcome) - neuropsychologial assessment by trained researcher
  comparison between follow up and baseline scores in neuropschological evaluations performed by specialist using SuperLab tool

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, PhD, Study Chair — Irmandade da Santa Casa de Misericórdia de São Paulo; Pedro Shiozawa, MD, Principal Investigator — Irmandade da Santa Casa de Misericóridia de São Paulo; Quirino Jr Cordeiro, PhD, Study Director — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (1):
- Centro de Atenção Integrada à Saúde Mental, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Loranger AW. Sex difference in age at onset of schizophrenia. Arch Gen Psychiatry. 1984 Feb;41(2):157-61. doi: 10.1001/archpsyc.1984.01790130053007. PMID 6696597
- [Background] Andrade L, Caraveo-Anduaga JJ, Berglund P, Bijl RV, De Graaf R, Vollebergh W, Dragomirecka E, Kohn R, Keller M, Kessler RC, Kawakami N, Kilic C, Offord D, Ustun TB, Wittchen HU. The epidemiology of major depressive episodes: results from the International Consortium of Psychiatric Epidemiology (ICPE) Surveys. Int J Methods Psychiatr Res. 2003;12(1):3-21. doi: 10.1002/mpr.138. PMID 12830306
- [Background] McGlashan TH, Johannessen JO. Early detection and intervention with schizophrenia: rationale. Schizophr Bull. 1996;22(2):201-22. doi: 10.1093/schbul/22.2.201. PMID 8782282
- [Background] Andreasen NC. Symptoms, signs, and diagnosis of schizophrenia. Lancet. 1995 Aug 19;346(8973):477-81. doi: 10.1016/s0140-6736(95)91325-4. No abstract available. PMID 7637483
- [Background] Bressan RA, Chaves AC, Pilowsky LS, Shirakawa I, Mari JJ. Depressive episodes in stable schizophrenia: critical evaluation of the DSM-IV and ICD-10 diagnostic criteria. Psychiatry Res. 2003 Jan 25;117(1):47-56. doi: 10.1016/s0165-1781(02)00298-6. PMID 12581820
- [Background] Bensenor IM, Brunoni AR, Pilan LA, Goulart AC, Busatto GF, Lotufo PA, Scazufca M, Menezes PR. Cardiovascular risk factors in patients with first-episode psychosis in Sao Paulo, Brazil. Gen Hosp Psychiatry. 2012 May-Jun;34(3):268-75. doi: 10.1016/j.genhosppsych.2011.12.010. Epub 2012 Feb 2. PMID 22305369
- [Background] Awad AG, Voruganti LN. The burden of schizophrenia on caregivers: a review. Pharmacoeconomics. 2008;26(2):149-62. doi: 10.2165/00019053-200826020-00005. PMID 18198934
- [Background] Brunoni AR, Teng CT, Correa C, Imamura M, Brasil-Neto JP, Boechat R, Rosa M, Caramelli P, Cohen R, Del Porto JA, Boggio PS, Fregni F. Neuromodulation approaches for the treatment of major depression: challenges and recommendations from a working group meeting. Arq Neuropsiquiatr. 2010 Jun;68(3):433-51. doi: 10.1590/s0004-282x2010000300021. PMID 20602051
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Davey NJ, Smith HC, Savic G, Maskill DW, Ellaway PH, Frankel HL. Comparison of input-output patterns in the corticospinal system of normal subjects and incomplete spinal cord injured patients. Exp Brain Res. 1999 Aug;127(4):382-90. doi: 10.1007/s002210050806. PMID 10480273
- [Background] Brunoni AR, Ferrucci R, Fregni F, Boggio PS, Priori A. Transcranial direct current stimulation for the treatment of major depressive disorder: a summary of preclinical, clinical and translational findings. Prog Neuropsychopharmacol Biol Psychiatry. 2012 Oct 1;39(1):9-16. doi: 10.1016/j.pnpbp.2012.05.016. Epub 2012 May 28. PMID 22651961
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710
- [Background] Wagner T, Fregni F, Fecteau S, Grodzinsky A, Zahn M, Pascual-Leone A. Transcranial direct current stimulation: a computer-based human model study. Neuroimage. 2007 Apr 15;35(3):1113-24. doi: 10.1016/j.neuroimage.2007.01.027. Epub 2007 Feb 4. PMID 17337213
- [Background] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793
- [Background] Fregni F, Pascual-Leone A. Technology insight: noninvasive brain stimulation in neurology-perspectives on the therapeutic potential of rTMS and tDCS. Nat Clin Pract Neurol. 2007 Jul;3(7):383-93. doi: 10.1038/ncpneuro0530. PMID 17611487